CLINICAL TRIAL: NCT04559672
Title: Cervical Laminoplasty Versus Laminectomy and Fusion: the Long-term Results Comparison
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Xuhua Lu, Director of Traumatic Orthopaedic Department, Shanghai Changzheng Hospital
Other Study IDs: CZ2020091101
Record Dates: First submitted 2020-09-13; First posted 2020-09-23 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Myelopathy Cervical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laminoplasty Group: Patients who underwent cervical laminoplasty surgery due to myelopathy.
  Interventions: Procedure: Cervical laminoplasty surgery
- Laminectomy and Fusion Group: Patients who underwent cervical laminectomy and fusion surgery due to myelopathy.
  Interventions: Procedure: Cervical laminectomy and fusion surgery

INTERVENTIONS:
Procedure: Cervical laminoplasty surgery — The posterior standard cervical laminoplasty procedure with ARCH mini-plate fixation
  Groups: Laminoplasty Group
Procedure: Cervical laminectomy and fusion surgery — The posterior standard cervical laminectomy and fusion surgery procedure with lateral mass screws fixation
  Groups: Laminectomy and Fusion Group

SUMMARY:
The objective of this study is to retrospectively analyze and compare the long-term clinical and radiographic results of multi-level laminoplasty to multi-level laminectomy and fusion for the treatment of patients with cervical myelopathy or myeloradiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years
* The patient has the diagnosis of degenerative cervical myelopathy
* The myelopathy or myeloradiculopathy requires a posterior cervical decompression of the spinal canal involving two or more contiguous intervertebral levels including and between C3 and C7
* More than five years of follow-up time

Exclusion Criteria:

* Presence of primary focal anterior compression of the cervical spinal cord
* Previous surgery of the cervical spine
* Tumor, infection, or trauma of the cervical spine or cord
* Patients with ankylosing spondylitis
* Patients with neurodegenerative diseases, or any neuropathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent cervical laminoplasty or laminectomy and fusion surgery due to degenerative cervical myelopathy in our hospital from January 1, 2005 to January 1, 2015 were screened and included according to the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of Japanese Orthopaedic Association Score (JOA) | baseline, 12 months post-treatment and through study completion, an average of 10 year
  Total score 0-17. The lower the score the more severe the deficits.
Change of Neck Disability Index (NDI) | baseline, 12 months post-treatment and through study completion, an average of 10 year
  Ranging from 0%-100%. A higher score indicates more patient-rated disability.
Change of Sagittal Lordosis Angle | baseline, 12 months post-treatment and through study completion, an average of 10 year
  Measured by lateral X-Ray image. The change of lordosis was calculated and compared.
Reoperation rate | through study completion, an average of 10 year
  Any reoperation involving the same segments or adjacent segments will be calculated.

SECONDARY OUTCOMES:
Change of Pain Scores on the Visual Analog Scale (VAS) | baseline, 12 months post-treatment and through study completion, an average of 10 year
  Ranging from 0-10. A higher score indicates more severe pain.
Change of Range of Motion | baseline, 12 months post-treatment and through study completion, an average of 10 year
  Measured by dynamic X-Ray image.
Complication rate | through study completion, an average of 10 year
  Any complications related to surgery will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Lu, M.D., Principal Investigator — Shanghai Changzheng Hospotal
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China